CLINICAL TRIAL: NCT04167280
Title: Regular Use Effect of Inhaled Ipratropium Bromide on Airway Responsiveness to Methacholine in Well-controlled Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Don Cockcroft, Professor, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Bio REB 1522
Record Dates: First submitted 2019-11-13; First posted 2019-11-18 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Asthma
Keywords: ipratropium bromide; methacholine PD20; tolerance
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ipratropium bromide (Active Comparator): 20mcg bronchodilator inhaler
  Interventions: Drug: Ipratropium Metered Dose Inhaler
- placebo (Placebo Comparator): matching bronchodilator inhaler
  Interventions: Drug: placebo metered dose inhaler

INTERVENTIONS:
Drug: Ipratropium Metered Dose Inhaler — MDI to deliver 20mcg per puff ipratropium bromide
  Arms: Ipratropium bromide
Drug: placebo metered dose inhaler — matched MDI to deliver inactive drug
  Arms: placebo

SUMMARY:
Study is looking at the development of tolerance to methacholine following regular use of ipratropium bromide in mild asthmatics.

DETAILED DESCRIPTION:
This study is being conducted people with well controlled (mild) asthma to determine if ipratropium bromide taken three times daily for six days (i.e. 2 puffs in the morning, 2 puffs in the afternoon and 2 puffs in the evening) followed by a final dose on the morning of day 7 reduces the effectiveness of this medication on blocking the effect of methacholine challenge.

ELIGIBILITY:
Inclusion Criteria:

* airway responsiveness to methacholine
* adequate baseline lung function
* no respiratory infection or exposure to stimuli that may alter response to methacholine within 4 weeks

Exclusion Criteria:

* pregnancy
* current smoker
* requirement for medications other than salbutamol that will interfere with airway response to methacholine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Methacholine PD20 | Pre treatment
  dose of methacholine required to induce a 20% fall in FEV1 (volume of air forcefully exhaled in one second)
Methacholine PD20 | Day 7 after starting treatment
  dose of methacholine required to induce a 20% fall in FEV1 (volume of air forcefully exhaled in one second)
Methacholine PD20 | 24 hours after last dose
  dose of methacholine required to induce a 20% fall in FEV1 (volume of air forcefully exhaled in one second)

CONTACTS AND LOCATIONS:
Overall Officials: Don Cockcroft, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No